CLINICAL TRIAL: NCT05024552
Title: A Phase 1 Study of Vyxeos Plus Gilteritinib in Relapsed or Refractory, FLT3-Mutated Acute Myeloid Leukemia
Brief Title: Vyxeos Plus Gilteritinib in Relapsed or Refractory, FLT3-Mutated AML
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20752
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia With FLT3/ITD Mutation
MeSH Terms: interventions — gilteritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Arm (Experimental): Participants will receive intravenous Vyxeos on days 1, 3 and 5 and Gilteritinib will be given on days 6-19 of induction therapy. The induction and reinduction dose of Vyxeos is 44mg/m2 daunorubicin and 100mg/m2 of cytarabine with each infusion.
  Dose level 1: Vyxeos + 120 mg Gilertinib
  In the event of a dose-limiting toxicity (DLT) at the initial dose level, a dose level minus (-) 1 is permitted Dose Level -1: Vyxeos + 80 mg Gilertinib
  Interventions: Drug: Gilteritinib; Drug: Vyxeos
- Dose Expansion Arm (Experimental): Participants will receive intravenous Vyxeos on days 1, 3 and 5 and Gilteritinib will be given on days 6-19 of induction therapy in the dose determined in the dose escalation arm.
  Interventions: Drug: Gilteritinib; Drug: Vyxeos

INTERVENTIONS:
Drug: Gilteritinib — Gilteritinib is an oral inhibitor of FLT3-ITD and FLT3-TKD. Dose cohort 1 will receive 120mg daily on days 6-19 of induction and days 4-17 of re-induction and consolidation
  Other Names: Xospata
Drug: Vyxeos — Vyxeos is a liposomal encapsulation of cytarabine and daunorubicin. It is given as an intravenous infusion over 90 minutes on days 1, 3 and 5 of induction and days 1 and 3 of re-induction and consolidation. The induction and reinduction dose is 44mg/m2 daunorubicin and 100mg/m2 of cytarabine with each infusion. The consolidation dose is 29mg/m2 daunorubicin and 65mg/m2 of cytarabine with each dose.
  Other Names: daunorubicin-cytarabine

SUMMARY:
This study combines vyxeos and gilteritinib in patients with relapsed or refractory FLT3-mutated acute myeloid leukemia. Vyxeos and gilteritinib will be given as induction therapy. Those patients entering a complete remission or a complete remission with incomplete blood count recovery will be allowed to proceed to consolidation therapy with vyxeos and gilteritinib. Those patients who do not proceed to an allogeneic stem cell transplant for any reason are able to enter the maintenance phase of this trial using daily gilteritinib

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* FLT3-ITD or FLT3-TKD mutated AML (non-M3) in 1st or greater relapse or refractory to at least one prior line of AML directed therapy
* FLT3 testing must be confirmed at the time of disease relapse
* Adequate organ function
* Left ventricular ejection fraction (LVEF) ≥50%
* Prior anthracycline exposure ≤368 mg/m2 daunorubicin (or equivalent)
* Ability to take oral medication and willingness to adhere to the medication regimen
* For females of reproductive potential: use of highly effective contraception including double barrier methods (condoms with spermicidal jelly or foam and diaphragm with spermicidal jelly or foam), oral, depo provera, or injectable contraceptives, intrauterine devices and tubal ligation.
* For females of reproductive potential: negative serum or urine pregnancy test with a sensitivity of at least 50mIU/mL within 10 days and again within 24 hours of beginning study treatment
* For males of reproductive potential: use of condoms
* Breastfeeding mothers must agree to discontinue nursing
* Patients who have relapsed after and allogeneic stem cell transplant must have controlled grade ≤2 GVHD. Immunosuppression with tacrolimus or sirolimus is allowed at stable or tapering doses.

Exclusion Criteria:

* Patients may not be receiving any other investigational agents
* Patients with documented central nervous system involvement of AML
* Progression of AML while on prior gilteritinib therapy
* Patients must not have evidence of GI tract abnormalities that would alter the absorption of oral medications
* Major surgery within two weeks of first dose of study drug. Patients must have recovered from the effects of any surgery performed greater than two weeks prior
* WBC count ≥50,000 at the time study treatment begins. Use of hydroxyurea to maintain WBC <50,000 is allowed up to the time that study treatment begins
* Predicted inability to tolerate standard induction chemotherapy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* No other malignancies in addition to AML that are currently requiring treatment with the exception of: 1) basal cell or squamous cell carcinoma or the skin; 2) carcinoma in situ of the cervix or breast; 3) a history of breast cancer that is currently being managed with adjuvant endocrine therapy
* Grade ≥3 acute or chronic graft versus host disease after allogeneic stem cell transplant. No steroids for GVHD are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-02-25 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Up to 18 months
  Dose escalation will determine the Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of Vyxeos plus Gilteritinib. The MTD is the highest dose of the combination therapy that dose not cause unacceptable side effects.

SECONDARY OUTCOMES:
Complete Remission Rate | Up to 18 months
  Rate of complete remission (CR) and complete remission with incomplete blood count recovery (CRi). The definition of CR and CRi is based on the European LeukemiaNet 2017 Response Criteria
Event free survival (EFS) | Up to 18 months
  Event free survival is determined as the duration of time from start of treatment to the time of cancer recurrence.
Overall survival (OS) | Up to 5 years
  Overall survival is defined as the duration of time from start of treatment to the time of death from any cause or date of last contact.

CONTACTS AND LOCATIONS:
Overall Officials: Onyee Chan, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://www.moffitt.org/clinicaltrialssearch/?diseasesite=&query=20752&studytype=&medication=&therapy=&pi=&nct=&sortcriteria=